CLINICAL TRIAL: NCT06505655
Title: Early Diagnosis of Acute Renal Failure, Which May Occur in Patients After Surgeries Requiring Hypotensive Anesthesia, by Urine Trehalase Levels.
Brief Title: Early Diagnosis of Acute Renal Failure by Urine Trehalase Levels.
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Istinye University
Other Study IDs: istinye university trehalase
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Trehalase Levels; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: trehalase levels — We think that in surgical patients requiring hypotensive anesthesia, acute kidney injury, which may occur due to intraoperative renal hypoperfusion, can be diagnosed early by evaluating the urine trehalase value using the ELISA method

SUMMARY:
We think that in surgical patients requiring hypotensive anesthesia, acute kidney injury, which may occur due to intraoperative renal hypoperfusion, can be diagnosed early by evaluating the urine trehalase value using the ELISA method, and thus, early diagnosed acute renal failure can be treated quickly and patients can be protected from subsequent complications in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18 and under the age of 65
* Having signed the BGOF form to be included in the study,
* Being in ASA 1 or ASA 2 classification
* Not having kidney failure or kidney disease
* No history of single kidney or renal transplantation
* Not using nephrotoxic drugs or agents before surgery
* Renal function tests taken preoperatively should be within normal ranges.
* No urinary tract infection or urinary problems (such as polyuria, oliguria or anuria)

Exclusion Criteria:

* Those under the age of 18 or over the age of 65
* Those who do not want to participate in the study
* ASA 3 and above
* Having previously received treatment for kidney disease - including kidney stones -
* Having been previously diagnosed with acute or chronic renal failure
* Having a single kidney or a history of renal transplantation
* Using nephrotoxic drugs or agents (such as contrast material) before surgery
* Kidney function tests taken preoperatively are not within normal ranges
* Having a urinary tract infection or urinary problem (such as polyuria, oliguria or anuria)
* Having a history of kidney stones, acute renal failure or chronic renal failure
* Those with active infection or disease before surgery
* They were determined as patients for whom consent was not obtained for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients between the ages of 18-65 who underwent a surgical operation requiring hypotensive anesthesia will be included in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
trehalase levels | 1 month
  urine trehalase levels

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chavan S, Hase N, Chavan P. Urinary enzymes in nephrotic syndrome. Indian J Clin Biochem. 2005 Jul;20(2):126-30. doi: 10.1007/BF02867411. PMID 23105544
- [Background] Ouyang Y, Xu Q, Mitsui K, Motizuki M, Xu Z. Human trehalase is a stress responsive protein in Saccharomyces cerevisiae. Biochem Biophys Res Commun. 2009 Feb 6;379(2):621-5. doi: 10.1016/j.bbrc.2008.12.134. Epub 2009 Jan 4. PMID 19126402
- [Result] Sasai-Takedatsu M, Kojima T, Taketani S, Ono A, Kitamura N, Kobayashi Y. Urinary trehalase activity is a useful marker of renal proximal tubular damage in newborn infants. Nephron. 1995;70(4):443-8. doi: 10.1159/000188643. PMID 7477650
- [Result] Sasai-Takedatsu M, Taketani S, Nagata N, Furukawa T, Tokunaga R, Kojima T, Kobayashi Y. Human trehalase: characterization, localization, and its increase in urine by renal proximal tubular damage. Nephron. 1996;73(2):179-85. doi: 10.1159/000189037. PMID 8773341